CLINICAL TRIAL: NCT02878577
Title: Monitoring Alterations Following Traumatic Brain Injury Using Clinical Evaluation, Neuropsychological Assessments, Structural and Functional MRI and EEG Analysis
Brief Title: Monitoring the Alterations That Occur in the Brain Following Traumatic Brain Injury
Acronym: TBI
Status: Completed | Type: Observational
Sponsor: ElMindA Ltd (Industry)
Collaborators: Sheba Medical Center (Other Government); Tel Aviv University (Other)
Responsible Party: Sponsor
Other Study IDs: ELM-37
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2019-01-04 (Actual); Status verified 2018-01

CONDITIONS: Traumatic Brain Injury (TBI)
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Magnetic Resonance Imaging; Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EEG fMRI TBI Mild/Moderate-Severe severity: patient population who suffered a brain trauma (traumatic brain injury, TBI). with a Glasgow Coma Scale between 3-15
  Interventions: Device: fMRI
- EEG fMRI Control group: healthy subjects with out a traumatic brain injury
  Interventions: Device: fMRI

INTERVENTIONS:
Device: fMRI — fMRI scans, mapping brain connectivity using EEG in combination with eye-tracking technology (Brain Network Activation (BNA) technology developed by ELMINDA), characterizing of cortical layers using magnetic resonance (the CoLI technology developed by Tel-Aviv University), and Diffusion Tensor Imaging (DTI) imaging (imaging of brain tracks).
  Other Names: EEG; CANTAB (computerized cognitive assessments)

SUMMARY:
This project, will combine the data collected from existing and innovative technologies: fMRI scans, mapping brain connectivity using EEG in combination with eye-tracking technology (the BNA technology developed by ELMINDA), characterizing of cortical layers using magnetic resonance (the CoLI technology developed by Tel-Aviv University), and DTI imaging (imaging of brain tracks). To do so, Sheba's Medical Center, Tel Hashomer, joined the project and is responsible for recruiting patients from the Department of Neurosurgery and Department of Rehabilitation and also is responsible for performing the needed tests.

DETAILED DESCRIPTION:
This research project is the continuation of the NOFAR project, collaboration between ELMINDA and Tel-Aviv University, which included a proof of concept of the technology developed in the university to characterize cortical layers using magnetic resonance. In light of the promising results, the partners have decided to make another leap forward, and test the technology amongst specific patient population who suffered a brain trauma (traumatic brain injury, TBI).

Early and proper diagnosis of brain injury is critical, since it can prevent further complications to the patient's health. The tests that are currently available are limited in their ability to provide a comprehensive and accurate assessment of the injured brain: imaging exams such as CT, MRI and PET help identify the location and severity of the injury but cannot provide data on the cognitive and functional effects of the injury. On the other hand, neuropsychological tests only allow examination of current cognitive functioning, and cognitive decline quantification is done according to mathematical models and subjective assessments of the patient and his family. Therefore, this area is lacking and it is important to find an objective measure that enables quantification of brain injury that will be an indication of cognitive decline.

The current project, will last two years, and will combine the data collected from existing and innovative technologies: fMRI scans, mapping brain connectivity using EEG in combination with eye-tracking technology (the BNA technology developed by ELMINDA), characterizing of cortical layers using magnetic resonance (the CoLI technology developed by Tel-Aviv University), and DTI imaging (imaging of brain tracks). To do so, Sheba's Medical Center, Tel Hashomer, joined the project and is responsible for recruiting patients from the Department of Neurosurgery and Department of Rehabilitation and also is responsible for performing the needed tests.

The product that will be developed at the end of the Magneton project is expected to be a unique analysis method that allows examination and monitoring of the affected brain in both a functional and anatomically-structural ultra-high resolution.

ELIGIBILITY:
Inclusion Criteria:

1. Had the Glasgow coma scale score of 3-15 after the incident. (group 1)
2. males and females Age: 18-60 (not during their military service).

Exclusion Criteria:

* History of neurological disorders, mental retardation or a previous head injury.
* Current diagnosis or history of psychiatric disorders.
* Drugs and / or alcohol dependence or abuse existed prior to the head injury.
* Unconsciousness.
* Pregnancy.
* Artificial respiration.
* Renal failure.
* Cardiovascular instability.
* Metabolic instability (water, electrolytes, sugar).
* Fever or evidence of microbiological pollutant.
* Uncontrolled seizures.
* Hydrocephalus.
* Patients with open wounds that are not bandaged, preventing the use of the EEG cap.
* Deafness or blindness.
* History of drugs that affect the nervous system in the 3 months prior to the injury.
* Inability to cooperate in carrying out the necessary tests

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: study population will include two groups of subjects: group 1: subjects after a traumatic brain injury group 2: control group
Sampling Method: Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2016-09-21 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-07-18 (Actual)

PRIMARY OUTCOMES:
fMRI responses to a cognitive executive task | 12 months
  measure Blood oxygen dependent signal (BOLD) response in exposure to RAVEN's progressive matrices during fMRI scan, the difference in responses between the groups (severe TBI, mild TBI, healthy subjects), and the longitudinal change (in course of a year).
MRI Structural changes | 12 months
  Using MRI scan and special protocols (DTI, COLI), The investigators will examine the difference between the groups (severe TBI, mild TBI, healthy subjects), and the longitudinal change (in course of a year).
EEG responses to cognitive tasks in combination of an eye-tracking method | 12 months
  The investigators will examine the difference in responses between the groups (severe TBI, mild TBI, healthy subjects), and the longitudinal change (in course of a year).
Cognitive scores on CANTAB (computerized cognitive assessments) | 12 months
  The investigators will examine the difference in responses to different cognitive exams between the groups (severe TBI, mild TBI, healthy subjects), and the longitudinal change (in course of a year).

SECONDARY OUTCOMES:
Correlations between the different methods | 12 months
  Correlations between the different methods - structural scans, functional scans, EEG, cognitive tasks, self-reported symptoms questionnaires and doctor's report.

CONTACTS AND LOCATIONS:
Overall Officials: Ofer Keren, MD, Principal Investigator — Shebe Academic Medical Center
Locations (1):
- The Chaim Sheba Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No